CLINICAL TRIAL: NCT00610935
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intramuscular Peramivir in Subjects With Uncomplicated Acute Influenza.
Brief Title: Intramuscular Peramivir in Subjects With Uncomplicated Acute Influenza
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated for administrative reasons.
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCX1812 311; HHS # O100200700032C (Registry Identifier: U.S. Department of Health & Human Services)
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Influenza
Keywords: Influenza; Subjects with uncomplicated acute influenza
MeSH Terms: conditions — Influenza, Human | interventions — peramivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo intramuscular injection
  Interventions: Drug: Placebo
- Peramivir (Experimental): Single intramuscular injection of 300mg peramivir
  Interventions: Drug: Peramivir

INTERVENTIONS:
Drug: Peramivir — To evaluate the efficacy of peramivir administered intramuscularly compared to placebo on the time to alleviation of clinical symptoms in adult subjects with uncomplicated acute influenza.
  Arms: Peramivir
Drug: Placebo — Single intramuscular injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and effectivess of a single intramuscular injection of peramivir for the treatment of subjects with acute, uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects age ≥18 years.
* A positive Influenza A and/or B Rapid Antigen Test (RAT) performed with a commercially available test kit on an adequate anterior nasal specimen, in accordance with the manufacturer's instructions. A negative initial RAT should be repeated within one-hour.
* Presence of fever at time of screening of ≥38.0 ºC (≥100.4 ºF) taken orally, or ≥38.5 ºC (≥101.2 ºF) taken rectally. A subject self-report of a history of fever or feverishness within the 24 hours prior to screening will also qualify for enrollment in the absence of documented fever at the time of screening.
* Presence of at least one respiratory symptom (cough, sore throat, or nasal symptoms) of at least moderate severity.
* Presence of at least one constitutional symptom (myalgia [aches and pains], headache, feverishness, or fatigue) of at least moderate severity.
* Onset of symptoms no more than 48 hours before presentation for screening.
* Written informed consent.

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Presence of clinically significant signs of acute respiratory distress.
* History of severe chronic obstructive pulmonary disease (COPD) or severe persistent asthma (See section 15.2).
* History of congestive heart failure requiring daily pharmacotherapy with symptoms consistent with New York Heart Association Class III or IV functional status within the past 12 months.
* Screening ECG which suggests acute ischemia or presence of medically significant dysrhythmia.
* History of chronic renal impairment requiring hemodialysis and/or known or suspected to have moderate or severe renal impairment (actual or estimated creatinine clearance <50 mL/min).
* Clinical evidence of worsening of any chronic medical condition (temporally associated with the onset of symptoms of influenza) which, in the investigator's opinion, indicates that such finding(s) could represent complications of influenza.
* Current clinical evidence, including clinical signs and/or symptoms consistent with otitis, bronchitis, sinusitis and/or pneumonia, or active bacterial infection at any body site that requires therapy with oral or systemic antibiotics.
* Presence of immunocompromised status due to chronic illness, previous organ transplant, or use of immunosuppressive medical therapy which would include oral or systemic treatment with > 10 mg prednisone or equivalent on a daily basis within 30 days of screening.
* Currently receiving treatment for viral hepatitis B or viral hepatitis C.
* Presence of known HIV infection with a CD4 count <350 cell/mm3.
* Current therapy with oral warfarin or other systemic anticoagulant.
* Receipt of any doses of rimantadine, amantadine, zanamivir, or oseltamivir in the 7 days prior to screening.
* Immunized against influenza with live attenuated virus vaccine (FluMist®) in the previous 21 days.
* Immunized against influenza with inactivated virus vaccine within the previous 14 days.
* Receipt of any intramuscular injection within the previous 14 days.
* History of alcohol abuse or drug addiction within 1 year prior to admission in the study.
* Participation in a previous study of intramuscular or intravenous peramivir or previous participation in this study.
* Participation in a study of any investigational drug or device within the last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (95):
  - Physical Express, Millbrook, Alabama
  - Alabama Family Medical Center, Tuscaloosa, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Clopton Clinic, Jonesboro, Arkansas
  - Research Solutions, LLC, Jonesboro, Arkansas
  - Kevin Adkins, MD, Mountain Home, Arkansas
  - NuLife Clinical Research, Inc., Anaheim, California
  - Impact Clinical Trials, Beverly Hills, California
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - Med Investigations Incorporated, Fair Oaks, California
  - Universal Biopharma Research Institute Inc., Fresno, California
  - Research Center of Fresno, Inc, Fresno, California
  - Harmony Clinical, Inc., Garden Grove, California
  - Allergy, Asthma, and Respiratory Care Medical Center, Long Beach, California
  - National Institute of Clinical Research, Los Angeles, California
  - Center for Clinical Trials, LLC, Paramount, California
  - San Diego Sports Medicine and Family Health Center, San Diego, California
  - Coastal Medical Research Group, Inc., San Luis Obispo, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Clinicos, LLC, Colorado Springs, Colorado
  - Longmont Clinic, P.C., Longmont, Colorado
  - Florida Research Network, LLC, Gainesville, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Eastern Research, Hialeah, Florida
  - Century Clinical Research Inc, Holly Hill, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Office of Roger J. Miller, Jr., MD, Jacksonville, Florida
  - MD Now Medical Center, Lake Worth, Florida
  - DMI Healthcare Group, Largo, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Compass Research LLC, Orlando, Florida
  - Pines Research, LLC, Pembroke Pines, Florida
  - Wilker/Powers Center for Clinical Studies, Saint Cloud, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Sandersville Family Practice Center, Sandersville, Georgia
  - Quincy Medical Group, Quincy, Illinois
  - Investigators Research Group, LLC, Indianapolis, Indiana
  - Welborn Clinic Gateway, Newburgh, Indiana
  - Medical Associates Clinic PC, Dubuque, Iowa
  - Heart of America Research Institute, Shawnee Mission, Kansas
  - American Medical Exams, P.A., Topeka, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Lung Clinic, Hazard, Kentucky
  - Winchester, Patton, Burgess, PSC, Whitley City, Kentucky
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Gulf Coast Research LLC, Lafayette, Louisiana
  - Byron Jackson, Shreveport, Louisiana
  - Professional Clinical Research-Benzonia, Benzonia, Michigan
  - Professional Clinical Research, Inc., Cadillac, Michigan
  - Professional Clinical Research-Interlochen, Interlochen, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Clinvest, Springfield, Missouri
  - Clinical Research Department, Bozeman, Montana
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Prarie Fields Family Medicine, P.C, Fremont, Nebraska
  - Quick Care Medical, Hamilton, New Jersey
  - Health Sciences Research Center at Asthma & Allergy Associates P.C., Elmira, New York
  - Health Sciences Research Center, Ithaca, New York
  - American Institute of Healthcare & Fitness, Raleigh, North Carolina
  - Community Medical Partners, Canfield, Ohio
  - Parsons Avenue Medical Clinic, Columbus, Ohio
  - Ohio Clinical Research LLC, Lyndhurst, Ohio
  - Physician Care PM, Edmond, Oklahoma
  - Urgent Care of Green County, Owasso, Oklahoma
  - Integrated Medical Research PC, Ashland, Oregon
  - Primary Physicians Research Inc., Pittsburgh, Pennsylvania
  - Warminster Medical Associates, PC, Warminster, Pennsylvania
  - New England Center for Clinical Research, Inc., Cranston, Rhode Island
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Paris View Family Practice, Greenville, South Carolina
  - Andras Koser, Greenville, South Carolina
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Holston Medical Group, PC, Bristol, Tennessee
  - Holston Medical Group, P.C., Kingsport, Tennessee
  - DiscoveResearch Inc., Beaumont, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - Intrinsic Research Data, Inc., Corpus Christi, Texas
  - Allergy/Immunology Research Center of North Texas, Dallas, Texas
  - Research Across America, Dallas, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - Dynamed Clinical Research, L.P., Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - GSA Research, San Antonio, Texas
  - San Antonio Preventive and Diagnostic Medicine, San Antonio, Texas
  - Optimum Clinical Research, Salt Lake City, Utah
  - J. Lewis Research Inc, Salt Lake City, Utah
  - J. Lewis Research Inc. Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc., Salt Lake City, Utah
  - Physicians Research Options, LLC, Saratoga Springs, Utah
  - J. Lewis Research Inc. FirstMed, West Jordan, Utah
  - Virginia Adult & Pediatric Allergy & Asthma, P.C Department of Clinical Research, Richmond, Virginia
  - Holston Medical Group, Weber City, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were centrally randomized in a ratio of 2:1 to a single dose of IM peramivir 300 mg or placebo, in accordance with a computer-generated randomization schedule prepared by a non-study statistician. Each subject's assignment to treatment was stratified according to smoking status and RAT test for influenza A or B.
Period: Overall Study
Arm/Group | Placebo | Peramivir
Started | 25 | 57
ITTI Population (Intent to treat - infected (ITTI) population included all subjects who were randomized, received at least one injection of study drug, and had proven influenza infection by at least one of the following assessments performed on a Screening/Baseline sample: positive PCR assay or positive viral culture for Influenza A or B.) | 25 | 55
ITT Population (Intent to treat (ITT) population included all randomized subjects for whom data were analyzed in the respective randomized treatment groups. The ITT population = Safety Population) | 25 | 57
Completed | 24 | 54
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Sponsor Discontinuation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population included all randomized subjects for whom data were analyzed in the respective randomized treatment groups. The ITT population was the primary population for analyses of demography and subject accountability as well as safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Peramivir | Total
Number analyzed (Participants) | 25 | 57 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (8.86) | 32.6 (12.67) | 33.0 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 28 | 42
  Male | 11 | 29 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 4 | 6
  White | 15 | 41 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 9 | 15
Current Smoking Behavior at Randomization [Number; unit: participants]
  Smoker | 4 | 14 | 18
  Non-smoker | 21 | 43 | 64
Influenza PCR Results [Number; unit: participants]
  Negative | 0 | 2 | 2
  Influenza A (H1N1) | 5 | 16 | 21
  Influenza A (H3N2) | 15 | 33 | 48
  Influenza A (IND) | 1 | 0 | 1
  Influenza B | 4 | 6 | 10
  Influenza A and B | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Time to Alleviation of Clinical Signs and Symptoms of Influenza
Description: The primary efficacy endpoint was the time to alleviation of symptoms of influenza in subjects diagnosed with influenza, defined as the time from injection of study drug to the start of the time period when a subject had Alleviation of Symptoms. A subject had Alleviation of Symptoms if each of the seven symptoms of influenza (cough, sore throat, nasal obstruction, myalgia [aches and pains], headache, feverishness, and fatigue) as self-assessed and recorded in the subject diary were either absent or were present at no more than mild severity level and at this status for at least 21.5 hours (24 hours minus 10%). No statistical testing was performed.
Time Frame: Up to 14 days
Population: A total of 80 subjects met the criteria for inclusion in the ITTI population as defined by a positive PCR assay for influenza A or B from the nasopharyngeal specimen obtained prior to administration of study treatment. Seventy-nine of these were included in the primary efficacy analysis for whom data for time to symptom alleviation were available; There was insufficient data from one subject in the placebo group to enable determination of the Time to Alleviation of Symptoms.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Peramivir
Number analyzed (Participants) | 24 | 55
hours | 118.3 [81.3 to 175.5] | 103.9 [81.7 to 126.8]

2. Secondary Outcome: To Evaluate Changes in Influenza Virus Titer in Nasopharyngeal Samples in Response to Treatment.
Description: The change in influenza viral titers was defined as the time-weighted change from Baseline in log_10 tissue culture infective dose_50 (TCID50/mL) and was summarized for each treatment group. The differences between the treatment groups were planned to be evaluated using a Wilcoxon Rank Sum Test controlling for current smoking behavior. Specimens for virologic culture and determination of influenza virus TCID50/mL were obtained at interval visits after treatment. As the study was terminated prematurely, no statistical testing was performed on these data.
Time Frame: Change from baseline assessed on days 3, 5 and 9.
Population: The Intent To Treat Infected population (ITTI) population included all subjects who were randomized, received study drug, and had confirmed influenza A and/or B by primary viral culture or PCR.
Measure: Median (Full Range); unit: influenza viral titer - log10 TCID50/mL
Arm/Group | Placebo | Peramivir
Number analyzed (Participants) | 20 | 49
influenza viral titer - log10 TCID50/mL
  Baseline | 3.75 [1.75 to 5.00] | 3.75 [1.50 to 5.00]
  Day 3 - Change from baseline | -2.25 [-4.25 to -0.25] | -2.75 [-4.25 to 1.00]
  Day 5 - Change from baseline | -3.00 [-4.25 to -0.75] | -3.00 [-4.50 to -1.00]
  Day 9 - Change from baseline | -3.00 [-4.50 to -1.50] | -3.25 [-4.50 to -0.75]

ADVERSE EVENTS:
Time Frame: Reports of TEAEs were collected from the time of study drug administration through to the follow-up period ending on Day 14.
Arm/Group | Placebo | Peramivir
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/57
Other Adverse Events (participants affected / at risk) | 13/25 | 26/57
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Peramivir (N=57)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Ageusia (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4)
Syncope Vasovagal (Nervous system disorders) | 3 (3) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Urine Protein Present (Investigations) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated at the discretion of the Sponsor after 82 of the planned 600 subjects were enrolled. The reason for study termination was to allow the Sponsor to focus development efforts on a more concentrated formulation which would also allow evaluation of higher doses of peramivir administered intramuscularly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-08-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT00610935/Prot_SAP_000.pdf